CLINICAL TRIAL: NCT06959485
Title: Oxygen Therapy in Diabetic Kidney Disease and Its Effect on Proteinuria and Blood Glucose Level
Brief Title: Oxygen Therapy in Diabetic Kidney Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hodna Abdullah Ahmed, Resident of Internal medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Oxygen Therapy
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Active Comparator): About 20 patients suffering from Diabetic kidney disease and will be treated by exposing to early morning air for 60 minutes (Early morning air" refers to the fresh, cool air found during the early hours of the day, (it's around 5-7 am, just before or after sunrise).
  Interventions: Biological: Oxygen Therapy
- Group B (Active Comparator): About 20 patients suffering from Diabetic kidney disease and will be treated by exposing to oxygen by non- rebreather mask (We choose oxygen by non- rebreather mask and no other ways of oxygen delivery system because it is the only available cost effective and non-invasive oxygen delivery device that can provide high oxygen flow that is close enough to HBOT)
  Interventions: Biological: Oxygen Therapy
- Group C (Active Comparator): About 20 patients suffering from Diabetic kidney disease and will be treated by exposing to hyperbaric oxygen therapy in a hyperbaric chamber at 2.5 ATA (atmospheres absolute) for 60 minutes per session (we choose 2.5 ATA hyperbaric oxygen therapy in a hyperbaric chamber (atmospheres absolute) for 60 minutes per session.
  Interventions: Biological: Oxygen Therapy
- Group D (Active Comparator): About 20 patients suffering from Diabetic kidney disease and will receive standard diabetes and Diabetic kidney disease management
  Interventions: Biological: Oxygen Therapy

INTERVENTIONS:
Biological: Oxygen Therapy — 1. To evaluate the effect of oxygen therapy (hyperbaric oxygen and oxygen by non- rebreather mask) and early morning air on proteinuria in patients with diabetic kidney disease.
  2. To evaluate the effect of oxygen therapy (hyperbaric oxygen and oxygen by non- rebreather mask) and early morning air on glycated haemoglobin in patients with diabetic kidney disease.
  3. Comparing the effects of oxygen therapy (hyperbaric oxygen and oxygen by non- rebreather mask), early morning air exposure, and standard care on kidney function
  Other Names: Standard diabetes and CKD management

SUMMARY:
Diabetic kidney disease (DKD) is the most significant cause of end-stage kidney disease (ESKD). Albuminuria, evolving from microalbuminuria to nephrotic-range proteinuria, is a clinical hallmark of diabetic nephropathy (DN). It develops in about a third of diabetic patients and is considered an independent risk factor in the progression of DN and for all-cause mortality.

DETAILED DESCRIPTION:
According to the International Diabetes Federation's report, over 530 million people worldwide have diabetes . About one-third of diabetic patients develop diabetic nephropathy (DN) after the incubation period, which may last several years.

Diabetic kidney disease (DKD) is the most significant cause of end-stage kidney disease (ESKD). Albuminuria, evolving from microalbuminuria to nephrotic-range proteinuria, is a clinical hallmark of diabetic nephropathy (DN). It develops in about a third of diabetic patients and is considered an independent risk factor in the progression of DN and for all-cause mortality.

The management of diabetes includes lifestyle modifications, pharmacological interventions, and emerging therapies such as hyperbaric oxygen therapy (HBOT). It involves exposing patients to high levels of oxygen in a pressurized chamber, leading to various physiological effects .

HBOT increases the level of oxygen in tissues by complete saturation of haemoglobin and increasing the partial pressure of oxygen dissolved in plasma. This enables oxygen to diffuse into tissues compromised by acute inflammation and microvascular disease and dysfunction.

ELIGIBILITY:
Inclusion Criteria:

- Diabetic male and female patients aged > 18 yrs with diabetic kidney disease (eGFR 30-90 mL/min/1.73m² and proteinuria >300 mg/day)

Exclusion Criteria:

* Age < 18 yrs
* Cardiovascular disease (thorough assessment of the patient's medical history (symptoms suggestive of CVD (e.g., chest pain, shortness of breath, fatigue), family history of CVD and risk factors (e.g., hypertension, hyperlipidemia, smoking). Physical Examination including blood pressure measurement, auscultation of heart sounds and assessment of peripheral pulses. Additional Diagnostic Tests: Stress test (stress ECG and stress echocardiography): Evaluate cardiac function under stress, which can help detect coronary artery disease or other CVD.
* Chronic lung disease (COPD, pulmonary fibrosis …
* Other chronic disease affecting kidney function (lupus nephritis).
* Pregnancy or lactation.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
Improving of proteinuria in diabetic kidney disease | 6 months
  to estimate urinary albumin-to-creatinine ratio in patients suffering form diabetic kidney disease

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Anwar Thabet, Professor, Study Chair — Assiut University
Locations (1):
- Assuit University hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided